CLINICAL TRIAL: NCT01356953
Title: Effects of Exercise Intensity on 24-h Ambulatory Blood Pressure in Type 2 Diabetics
Brief Title: Exercise Intensity and Type 2 Diabetics
Acronym: EIT2D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of Brasília (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Pâmella Karoline de Morais, Universidade Católica de Brasília
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MORAIS0132008
Record Dates: First submitted 2011-05-10; First posted 2011-05-20 (Estimated); Last update posted 2011-05-20 (Estimated); Status verified 2008-09

CONDITIONS: Type 2 Diabetes
Keywords: Aerobic Exercise; Blood Pressure
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Aerobic Exercise (Experimental)
  Interventions: Other: Aerobic exercise

INTERVENTIONS:
Other: Aerobic exercise — Intensity of aerobic exercise

SUMMARY:
The purpose of this study is to determine if a single session of aerobic exercise effectively controls the blood pressure (BP) of individuals with type 2 diabetes mellitus (T2DM) over the 24h of post-exercise period, and the effects of intensity of aerobic exercise on these BP responses.

ELIGIBILITY:
Inclusion Criteria:

* sedentary
* a diagnosis of T2DM for at least one year
* glycemic control through nutrition and/or medication

Exclusion Criteria:

* be not under use of exogenous insulin and do not present chronic complications such as diabetic foot
* nephropathy
* retinopathy
* neuropathies and cardiovascular diseases

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-10; Primary Completion 2009-07 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Blood Pressure - Ambulatory blood pressure monitoring (ABPM) | Participants will be followed for the duration of experimental tests, an expected average of 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University of Brasilia, Taguatinga, Brazil